CLINICAL TRIAL: NCT01785940
Title: Evaluation of Ultrasound Guided Continuous Interscalene Block for Same Day Discharge Following Total Shoulder Arthroplasty - An Open Label Feasibility Study
Brief Title: Continuous Interscalene Block for Same Day Discharge Following Total Shoulder Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Shalini Dhir, Principal Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 103329
Record Dates: First submitted 2013-02-05; First posted 2013-02-07 (Estimated); Last update posted 2017-02-14 (Actual); Status verified 2017-02

CONDITIONS: Pain, Shoulder
Keywords: Interscalene Block; Perineural catheter; Ropivacaine; Postoperative pain; Home regional
MeSH Terms: conditions — Shoulder Pain; Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Interscalene block (Experimental): Interscalene catheters will be placed under aseptic precautions in each patient by one of the investigators using combined peripheral nerve stimulation and ultrasound guidance to get twitch in the C5-C6 dermatomes and documented spread of injectate near C5-6 nerve roots. Twenty mL of 0.2% ropivacaine will be injected while documenting adequate drug spread under ultrasound. After 20 min of injection, the interscalene nerve block will be evaluated and considered successful with inability to abduct the shoulder and a decrease in perceived sensation to cold of the skin over the deltoid muscle.
  Interventions: Procedure: Interscalene block

INTERVENTIONS:
Procedure: Interscalene block — Interscalene catheters will be placed under aseptic precautions in each patient by one of the investigators using combined peripheral nerve stimulation and ultrasound guidance to get twitch in the C5-C6 dermatomes and documented spread of injectate near C5-6 nerve roots. Twenty mL of 0.2% ropivacaine will be injected while documenting adequate drug spread under ultrasound. After 20 min of injection, the interscalene nerve block will be evaluated and considered successful with inability to abduct the shoulder and a decrease in perceived sensation to cold of the skin over the deltoid muscle.

SUMMARY:
Total shoulder surgeries are associated with considerable postoperative pain which may prevent rehabilitation and early discharge from the hospital. Continuous interscalene blocks with home infusions are commonly performed for pain relief following total shoulder arthroplasties. We want to evaluate the time to readiness for discharge following interscalene blocks in patients undergoing total shoulder arthroplasties.

DETAILED DESCRIPTION:
The number of shoulder replacement surgeries is increasing over the years and it is expected to continue as the population ages (1). This necessitates adequate pain control in the immediate and early postoperative period when pain levels are typically high. Adequate analgesia ensures patient comfort and the ability to perform physical therapy exercises associated with positive surgical outcomes (2-3). Interscalene brachial plexus block (ISB) is commonly performed to provide analgesia for patients undergoing surgical procedures in the shoulder region. Either single injection blocks or continuous perineural infusions are performed along with oral medications for better pain control in these patients. Compared with intravenous opioids, ISB is known to produce superior analgesia after major shoulder surgery (4,5). There are reports of outpatient TSA discharged directly from the recovery room following the use of continuous ISB but achievement of adequate range of motion were not tested in them (6). Consequently, ambulatory ISB may offer decreased hospitalization while ensuring adequate analgesia after TSA. Ilfeld et al (7) prospectively compared ISB and opioids regarding the time to readiness for discharge following TSA, which was followed by many other studies demonstrating the safety and efficacy of continuous ISB for TSA (8, 9). Ilfeld et al (6) showed that discharge criteria were 21 (16-41) h with the use of ISB as compared to 51 (37-90) h for those receiving perineural normal saline. In our centre, healthy patients requiring shoulder arthroplasty usually remain as in-patients for management of pain. Perineural infusions may be continued at home using a portable infusion pump after discharge. With the use of disposable portable infusion pump for continuous ISB, it may be feasible to discharge patients and reduce hospitalization time.

Although the study by Ilfeld et al showed continuous ISB allowing earlier home discharge following TSA, the patients in the study were evaluated for readiness to discharge on POD1 at 10 AM rather than the earliest times possible. Another interesting finding is that all patients received ropivacaine infusions till 6 AM of POD1 but the authors also claim to have discharged few patients on the same afternoon after the surgery. The block infusions reported in previous studies are higher than used at our institute.

There is also conflicting evidence that although continuous ISB provides adequate analgesia, they seldom impact early functional rehabilitation (10). With this background we want to evaluate the earliest times for the achievement of readiness to discharge with the use of ISB following TSA.

ELIGIBILITY:
Inclusion Criteria:

1. Male and females of 18-80 years of age, scheduled to undergo elective shoulder arthroplasty.
2. ASA Class I, II, III

Exclusion Criteria:

1. Patients with associated significant cardiac and respiratory disease.
2. Patients who will need hospitalization due to reason other than the planned surgery.
3. Patients with coexisting sleep apnea or morbid obesity (BMI> 35).
4. Patients with pre-existing major organ dysfunction such as hepatic and renal failure.
5. Psychiatric illnesses.
6. Lack of informed consent.
7. Allergy to any of the drugs used in the study.
8. Contraindications to interscalene block

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Pain scores: Visual analog scores | first 24 postoperative hours
  The patients will be evaluated for home discharge based on the degree of analgesia (VAS scores of < 40/100 on movement) at arrival to PACU, and at every 2 hours for the first 6 hours postoperatively and every 4 hourly till 6 AM on the morning of POD1 and at 23 postoperative hours.

SECONDARY OUTCOMES:
Range of motion | First 24 postoperative hours
  The patients will be evaluated for achievement and maintenance of at least 50% of expected range of motion at arrival to PACU, 6 hours postoperatively and on the morning of POD1 and at 23 postoperative hours.

OTHER OUTCOMES:
Analgesic consumption | First 24 postoperative hours
  Total analgesic consumption per day and the number of boluses used per day will be prospectively collected
Satisfaction score | 5th postoperative day
  Patient satisfaction will be documented on a visual analogue scale where 0 is totally dissatisfied and 100 is totally satisfied.
Readiness for home discharge | first 24 postoperative hours
  The time from the arrival in PACU to the attainment of home discharge criteria following exercises will be noted as the time to readiness for discharge.
Complication rates | first 5 postoperative days
  Adverse events such as local anesthetic toxicity, neurological deficits respiratory insufficiency will be prospectively collected. The failure rate and the number of attempts will also be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Shalini Dhir, FRCPC, Principal Investigator — St Joseph's Health Care centre, London, ontario
Locations (1):
- St. Joseph's Hospital, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ilfeld BM, Wright TW, Enneking FK, Mace JA, Shuster JJ, Spadoni EH, Chmielewski TL, Vandenborne K. Total shoulder arthroplasty as an outpatient procedure using ambulatory perineural local anesthetic infusion: a pilot feasibility study. Anesth Analg. 2005 Nov;101(5):1319-1322. doi: 10.1213/01.ANE.0000180199.52383.CE. PMID 16243987